CLINICAL TRIAL: NCT05958680
Title: ASDactive: Feasibility of An Integrated Theory-based Intervention to Promote Habitual Physical Activity Behaviours in Autistic Youth
Brief Title: ASDactive: An Integrated Theory-based Intervention to Promote Habitual Physical Activity
Acronym: ASDactive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aberystwyth University (Other)
Responsible Party: Principal Investigator, Kathrine Parsons, Principal Investigator, Aberystwyth University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20880
Record Dates: First submitted 2022-01-07; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Physical Inactivity; Sedentary Behavior; Autism; Autism Spectrum Disorder; Asperger Syndrome; Behavioral
Keywords: behavior change; physical activity; exercise; autism; aspergers; feasibility; implementation mapping
MeSH Terms: conditions — Sedentary Behavior; Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASDactive (Experimental): Theoretically derived behaviour change intervention aimed at promoting habitual physical activity uptake
  Interventions: Behavioral: ASDactive

INTERVENTIONS:
Behavioral: ASDactive — An integrated theory-based intervention to promote habitual physical activity behaviours in autistic youth

SUMMARY:
ASDactive is a theory-based behaviour change intervention aimed at improving the physical activity behaviours of autistic youth. The feasibility of the intervention will be tested through interviews with participants and stakeholders. "Proof of concept" will be tested through preliminary measures of physical activity measured before and after the intervention.

DETAILED DESCRIPTION:
ASDactive is has been developed with guidance from autistic people and stakeholders in autism. It is informed by motivation and behaviour change theory, specifically habit theory. The intervention aims to improve the habitual exercise behaviours of autistic youth by focusing on their strengths and interests.

The feasibility study will run for 3-months, with a further 3-month follow-up period. Participants will attend motivational sessions in person where they will self-select physical activity habits to incorporate into their daily lives. They will be taught fundamental movement skills that they can use in their own leisure time. In-person sessions will be held once per fortnight with online sessions twice weekly. Participants will be encouraged to engage with as many sessions as possible, but part of the evaluation will assess uptake and engagement.

Self-determination theory and habit theory will underpin all aspects of the intervention and autistic strong interests will be embedded in the materials used.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged 10-24-years diagnosed with Level 1 autism or Asperger's syndrome

Exclusion Criteria:

* Physical conditions or injuries that might hinder physical activity participation

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention through its Adoption | 3- months
  Number of people engaging with the sessions each week
Feasibility through Implementation | 3- months
  Assessment of the fidelity of the delivery sessions. Two sessions will be recorded and reviewed by two assessors to ensure they are consistently delivered according to the protocol

SECONDARY OUTCOMES:
Self-Report Habit Index | 3- and 6-months as a follow-up
  A scale which measures a combination of subjective estimates (never to always) and recall of behavioural frequency (number of times per week). These are then multiplied by stability of context measured by subjective evaluations (e.g., always in the same place to never in the same place). When frequency and stability are multiplied on the scale, a habit strength between 0-36 is given. Lower scores indicate poor levels of habit strength, higher scores indicated good habit strength.
Basic Psychological Need Satisfaction Scale | 3 months
  Measures of basic psychological needs (autonomy, relatedness, and competence) measured on a 7-point likert scale from strongly disagree to strongly agree. Lower scores indicate lower levels of perceived psychological needs being met and so worse outcomes.
International Physical Activity Questionnaire- Short form | 3- and -6 months as a follow-up
  self-report physical activity levels through open-ended questions surrounding individuals' last 7-day recall of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Parsons, Principal Investigator — Aberystwyth University
Locations (1):
- Katherine Parsons, Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD will be stored in Aberystwyth University's repository for 5-years. IPD will not include personal data belonging to participants but will include anonymised outcome data generated from self-report measures.
Supporting Information: Study Protocol, SAP
Time Frame: 5-years
Access Criteria: Access can be granted via Aberystwyth University